CLINICAL TRIAL: NCT02265874
Title: Nicotine Treatment for Pulmonary Sarcoidosis: A Clinical Trial Pilot Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Elliott Crouser, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2014H0291
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): Habitrol Nicotine patch - 7,14,21 mg patches Qd
  Interventions: Drug: Habitrol
- Control (Placebo Comparator): Placebo patch
  Interventions: Drug: Placebo to Habitrol

INTERVENTIONS:
Drug: Habitrol — Patch used daily for 28 weeks
  Arms: Treatment
Drug: Placebo to Habitrol
  Arms: Control

SUMMARY:
The purpose of this study is to determine if nicotine treatment is beneficial for the treatment of sarcoidosis. Sarcoidosis is a disease of unknown cause that leads to inflammation. This disease affects your body's organs.

DETAILED DESCRIPTION:
Participants will be randomly divided into two groups. One group will receive a nicotine patch to use for approximately 7 months; the other group will receive placebo for nicotine patches to use for the same time period.

Both groups will be contacted weekly by phone for the first 3 weeks then monthly for the duration of the study to monitor for any side effects.

The following information and samples will be collected:

Questionnaires Medical History Spirometry CT Scans Physical Exam Blood Samples for nicotine and nicotine metabolites

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects ≥ 18 to ≤ 75 years of age will be screened for eligibility.
* Eligible adult patients will have histologically proven sarcoidosis, diagnosed at least 6 months before screening, evidence of parenchymal disease on chest radiograph, an FVC between 50% and 85% of the predicted value, and a Medical Research Council dyspnea score (47) of at least grade 1.
* Patients must have been treated with at least 10 mg/day of prednisone or equivalent or one or more immunomodulating agents (hydroxychloroquine, methotrexate, azathioprine, leflunomide) for >3 months before screening.
* Doses of these medications must be stable for at least 1 month before study entry.
* During the study, background medication regimen and doses are to remain stable.

Exclusion Criteria:

* active tobacco smoking or use of smokeless tobacco products containing nicotine,
* active cardiac or central nervous system disease,
* history of adverse reaction to nicotine or nicotine-containing products,
* patients with extensive irreversible pulmonary fibrosis (based upon lung biopsy or high resolution CT scan criterion) or inability to provide consent.

The subject will be excluded if they have a smoking history of greater than 20 pack years, or a diagnosis of other significant respiratory disorder other, than sarcoidosis that, in the opinion of the investigator, would complicate the evaluation of response to treatment; or, history of substance abuse (drugs or alcohol) within 3 years prior to screening or other circumstances (e.g., psychiatric disease) that could interfere with the subject's adherence to protocol requirements or increase their risk of drug (nicotine) dependence.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10-21 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Martha Morehouse Medical Pavilion 2050 Kenny Rd; Ste 2600, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan in place to share IPD

REFERENCES:
- [Result] Crouser ED, Smith RM, Culver DA, Julian MW, Martin K, Baran J, Diaz C, Erdal BS, Hade EM. A Pilot Randomized Trial of Transdermal Nicotine for Pulmonary Sarcoidosis. Chest. 2021 Oct;160(4):1340-1349. doi: 10.1016/j.chest.2021.05.031. Epub 2021 May 23. PMID 34029565
- [Result] Hade EM, Smith RM, Culver DA, Crouser ED. Design, rationale, and baseline characteristics of a pilot randomized clinical trial of nicotine treatment for pulmonary sarcoidosis. Contemp Clin Trials Commun. 2020 Oct 7;20:100669. doi: 10.1016/j.conctc.2020.100669. eCollection 2020 Dec. PMID 33089005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2015 through January 2019 from The Ohio State University Medical Center and from Cleveland Clinic Foundation
Pre-assignment Details: Patients were screened for lung fibrosis and for cardiac involvement of sarcoidosis and were excluded if these were present
Groups:
- Habitrol: Habitrol Nicotine patch - 7,14,21 mg patches Qd
  Habitrol: Patch used daily for 28 weeks
- Placebo: Placebo patch - 7,14,21 mg patches Qd
  Placebo to Habitrol
Period: Overall Study
Arm/Group | Habitrol | Placebo
Started | 24 | 26
Completed | 20 | 20
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Habitrol | Placebo | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (11.5) | 55.8 (8.0) | 53.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 18 | 16 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Forced Vital Capacity (FVC)
Description: changes in forced vital capacity (FVC) measured by pulmonary function testing (breathing tests) measured in liters
Time Frame: 28 weeks
Population: Change in FVC from baseline to week 28 (study completion) in Habitrol treatment group compared to Placebo treatment group.
Measure: Mean (Standard Error); unit: liters
Groups:
- Control: Placebo patch
  Placebo to Habitrol
Arm/Group | Treatment | Control
Number analyzed (Participants) | 20 | 20
liters | 0.07 (0.22) | -0.07 (0.04)

2. Secondary Outcome: Changes Detected by Computed Tomography (CT) of Lungs
Description: CT lung scans are analyzed by a computer program: Briefly, lung architecture, manifest as pixelated Houndsfield units, is assessed for regional mismatches (texture), wherein linear conformation of pixels are removed (equating with airways, blood or lymphatic vessels) and the mismatched pixels are quantified (i.e., Lung Texture Score; LTS) and are reflective of lung anatomy, including lung nodules, interstitial fibrosis or alveolar ground glass (i.e., pulmonary sarcoidosis manifestations). LTS is represented by arbitrary units, and are reported to range from 25 - 70; 25-40 being within the normal range (i.e., normal lung anatomy; and values in the 40 - 70 range are associated lung parenchymal disease (PMID: 22628482).
Time Frame: 28 weeks
Population: Change in lung texture score from baseline to study completion in the Habitrol treatment group compared to the Placebo group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 20 | 20
score on a scale | -1.0 (3.5) | 2.5 (3.5)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded over a period of 6 months for each participant
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 6/24 | 2/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=24) | Control (N=26)
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 2 (2) — Headache without neurological impairment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT02265874/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT02265874/ICF_001.pdf